CLINICAL TRIAL: NCT04174404
Title: Developing and Testing the Effectiveness of Intelligent Customer-driven Solution for Pediatric Surgery Care on the Improvement of Outcomes of Parents and Their Children Undergoing Circumcision
Brief Title: Intelligent Customer-driven Solution for Pediatric Surgery Care for Parents and Their Children Undergoing Circumcision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HE Hong-Gu (Other)
Collaborators: National University Hospital, Singapore (Other); Buddy Healthcare Ltd OY (Unknown)
Responsible Party: Sponsor-Investigator, HE Hong-Gu, Associate Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2019/00582
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Circumlocution; Children; Surgery; Parents
Keywords: Pediatric Surgery Care; Circumcision; Children; Parent; perioperative care; randomised controlled trial; Self-efficacy; Preoperative anxiety

STUDY DESIGN:
Intervention Model Description: This study will be a two-group pretest and repeated posttest pilot randomised controlled trial followed by a qualitative process evaluation. A randomized controlled trial design was chosen as it has been the gold standard in testing effectiveness of a new intervention or treatment. A qualitative process evaluation is incorporated into this study design to explore the experiences of the participants' use of the applications.
  A total of 80 dyads of parents and their primary school-aged children (7-12 years old) will be randomly assigned into the intervention group which will receive the ICory-Circumcision plus routine care, whereby the parents will receive the BuddyCare application while the child will receive the Triumf game application, and the control group, who will just receive routine care provided by the hospital.
Who Masked: Outcomes Assessor
Masking Description: The investigators will firstly generate certain sets of random numbers from 1 to 6 by using Research Randomiser (Research Randomiser, 2019). Each number represents one combination of the allocations, e.g. 1 - [I I C C}, 2 - {I C I C}, 3 - {I C C I}, 4- {C I C I}, 5- {C I I C} and 6 - {C C I I} where I and C represent the allocation to the intervention and control group, respectively. Such randomly generated sequences will be used to allocate participants, who will be assigned in successive order according to the sequence. Opaque, sealed envelopes with cardboard inside indicating the randomly assigned group will be prepared by the PI. Through these processes, randomisation and allocation concealment will be ensured (Doig & Simpson, 2005; Schulz & Grimes, 2002).
  One research assistant will recruit participant, collect baseline data, conduct randomisation, and deliver the intervention, while another research assistant who is blind from group allocation will collect post-test data.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in the intervention group will receive the routine care plus the ICory-Circumcision which is specially developed for this study based on preliminary studies, other literature, and most importantly, the surgical pathway currently practiced in the study hospital. The ICory-Circumcision programme has two components: (1) the Buddy Healthcare mobile app (BuddyCare) that provides a comprehensive day-by-day perioperative guide for parents regarding their child's surgery with an interface for health care professionals to monitor parents' and their children's needs as well as communicate with them. (2) The Triumf Health mobile game app that provides emotional support and distraction to children.
  Interventions: Other: ICory-Circumcision; Other: Routine care
- Control group (Active Comparator): The participants in the control group will receive routine care provided by the hospital which consists of normal doctor consultant, preoperative preparation, and postoperative care.
  Interventions: Other: Routine care

INTERVENTIONS:
Other: ICory-Circumcision — The ICory-Circumcision is specially developed for this study based on preliminary studies, other literature, and most importantly, the surgical pathway currently practiced in the study hospital. The ICory-Circumcision programme has two components: (1) the Buddy Healthcare mobile app (BuddyCare) that provides a comprehensive day-by-day perioperative guide for parents regarding their child's surgery with an interface for health care professionals to monitor parents' and their children's needs as well as communicate with them. (2) The Triumf Health mobile game app that provides emotional support and distraction to children. The ICory-Circumcision programme is designed to be a self-guided and healthcare professional-led. Participants will have access to BuddyCare for parents and Triumf Health from time of recruitment till 2 weeks after surgery while the healthcare professional would receive face-to-face training on how to use the BuddyCare dashboard.
  Arms: Intervention group
Other: Routine care — The routine care consists of normal consultations with the doctor, preoperative preparation, and post-operative care. During the first consultation, the child will be assessed for the need for circumcision and the doctor explains verbally to the parents about the procedure, risks, what to expect and prepare pre-operatively.

SUMMARY:
This study aims to (1) develop an intelligent customer-driven solution for pediatric surgery care for parents of children undergoing circumcision and their children; (2) examine the effectiveness of the intervention on outcomes of parents (self-efficacy in child care, perioperative knowledge, and satisfaction in perioperative care, need for information and anxiety) and children (preoperative anxiety and postoperative pain); and (3) explore users' (parents, children, health care professionals) perceptions of the intervention and suggestions for improvement.

DETAILED DESCRIPTION:
Objectives: The aims of this study are: (1) to develop an intelligent customer-driven solution for pediatric surgery care for parents of children undergoing circumcision (ICory- Circumcision) and their children; (2) to examine the effectiveness of the ICory- Circumcision on outcomes of parents (self-efficacy in child care, perioperative knowledge, and satisfaction in perioperative care, need for information and anxiety) and children (preoperative anxiety and postoperative pain), as well as no-show/ delayed show up for operation cases and health services use; and (3) to explore users' (parents, children, health care professionals) perceptions of the intervention and suggestions for improvement.

Study design: This study will be a two-group pretest and repeated posttest pilot randomised controlled trial followed by qualitative process evaluation. A total of 80 dyads of parents and their primary school-aged children (7-12 years old) will be randomly assigned into the intervention group which will receive the ICory-Circumcision plus routine care, whereby the parents will receive the BuddyCare application while the child will receive the Triumf game application, and the control group, who will just receive routine care provided by the hospital. An interview guide will be developed and used to interview the parents and healthcare professionals who used ICory-Circumcision to explore their experiences and opinions on strengths, weaknesses and areas for improvement. The children who have used the Triumf game will also be interviewed to explore their experiences about the game application.

Hypothesis: When compared to the control group, (1) parents in the intervention group who receive the ICory-Circumcision will report a significantly (a) higher level of self-efficacy in child care; perioperative knowledge and satisfaction (b) lower level of needs for information and preoperative anxiety. (2) The children in the intervention group will report a significantly lower level of preoperative anxiety and postoperative pain. (3) The intervention group will have fewer cases of no-show/ delayed show up for operation, and reduced health services use (e.g. reduced A & E department or GP attendance for non-medical reasons) within 2 weeks after the surgery.

ELIGIBILITY:
Children

Inclusion Criteria:

* age between 7-12 years old;
* is scheduled for an elective circumcision surgery;
* Is able to speak, and read in English;
* is accompanied by their parents (either mother or father or both) during the perioperative period; and
* has access to smart phone/tablet (own or rent from the project).

Exclusion Criteria:

* cognitive and learning disabilities identified from the medical record;
* a chronic illness and/or pain that required special medical care;
* anxiety disorder and other mood disorder as identified from their medical records;
* Hearing or visual impairments;
* depth perception deficits; and/or
* in the bereavement period in the past 6 months.

Parents

Inclusion Criteria:

* father or mother as main caregiver of the child who meet the aforementioned selection criteria;
* are 21 years and above;
* Able to communicate verbally and be literate in English; and
* have access to smart phone/tablets (own or rent from the project).

Exclusion Criteria:

* have visual/hearing impairment;
* have any cognitive impairment/mental disorder including anxiety disorder;
* have end stage of diseases; and/or
* in the bereavement period in the past 6 months.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Parents' preoperative anxiety and information requirement | Parents' preoperative anxiety and information requirement will be assessed at baseline (around 2 weeks before surgery) and will assess change between baseline and on the surgery day before the operation.
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS) (Moerman, van Dam, Muller & Oosting, 1996) will be used to measure parents' preoperative anxiety and information requirement. The APAIS is a six-item questionnaire consisting of 4 questions about the fear of anesthesia and procedure while 2 questions are about the need for information. The questionnaire is scored based on a likert scale of 1 to 5. A score of 1 would mean 'not at all' while 5 would mean 'extremely'. The total score for the anxiety scale can range from 4 to 20 while the need for information scale ranges from 2 to 10. The higher the scores, the higher the anxiety and the information required by the respondents.
Parents' perioperative knowledge | Parents' perioperative knowledge will be assessed at baseline (around 2 weeks before surgery) and will assess change between baseline and post-intervention at 2 weeks after surgery,
  The self-developed Parents' Perioperative Knowledge Questionnaire (PPKQ) will be used for assessing parents' perioperative knowledge with regards to the circumcision. It was developed by the study team. A content validity will be done by an expert panel consisting of 5-10 experts (Gilbert & Prion, 2016). The PPKQ contains 10 multiple choices questions. The higher number of questions answered correctly would indicate a higher understanding of the comprehension of the perioperative process thus better knowledge.
Parents' self-efficacy in child care | Parents' self-efficacy will be assessed at baseline (around 2 weeks before surgery) and will assess change between baseline and post-intervention at 2 weeks after surgery,
  A self-developed Parents' Self-Efficacy in Children's Perioperative Care (PSeCPC) questionnaire will be used to measure parents' self-efficacy in childcare throughout the perioperative process. There are 8 items for this scale and each item is rated on four responses: 1= not confident at alll, 2= a little confident, 3= moderately confident, 4=quite confident and 5= extremely confident. The total score is 8-40. Higher score means better self-efficacy.
Parents' satisfaction with Perioperative Care | Parents' satisfaction with Perioperative Care will be assessed at post-intervention around 2 weeks after surgery.
  A 6-point Ordinal Descriptive Scale - Satisfaction with Perioperative Care (ODS-SPC) will be used to assess parents' satisfaction with ICory-Circumcision and routine care. The scale only consists of one item and it is scored on a 6-point ordinal scale of 1 for "Very dissatisfied" to a score of 6 for "Very satisfied". The total score can range from 1 to 6. A higher score would indicate higher satisfaction with the perioperative care.
Children's preoperative anxiety: Modified Yale Preoperative Anxiety Scale - Short Form (mYPAS-SF) | Children's preoperative anxiety will be assessed on the day right before the operation.
  Modified Yale Preoperative Anxiety Scale - Short Form (mYPAS-SF) (Jenkins, Fortier, Kaplan, Mayes & Kain, 2014) will be used to measure the preoperative anxiety levels of the children right before the operation. It is a 4-item scale (activity, vocalization, emotional expressivity, state of apparent arousal) and it is filled in via observation. The total score ranges from 23 to 100. Higher scores mean higher levels of anxiety. A score of 31 and above would indicate high-anxiety (Kain et al., 1997; Rema, Cavaleiro, Pina & Machado, 2016).
Children's postoperative pain: The Faces Pain Scale | Children's postoperative pain will be measured at 24 hours post-surgery.
  The Faces Pain Scale - Revised (FPS-R) (International Association for the Study of Pain [IASP], 2001) will be used to assess the postoperative pain of the children. The FPS-R shows six faces with different facial expressions and the child is given instructions to point to the face corresponding to the amount of pain he feels at that moment. The scores range from 0-10 with a higher score means greater pain.
Health services use | Health services use will be assessed around 2 weeks after surgery.
  Health services use will be assessed by Healthcare Services Utilisation Questionnaire (HSUQ) to capture post-discharge information on resource utilization for each participant, e.g. emergency room attendance, and unplanned medical consultation at GP/ private clinic. The minimal service use will be zero, but there is no maximal limited. The higher value of services use indicates worse outcome.
Process evaluation | Process evaluation will be conducted around 2 weeks after surgery.
  Process evaluation will be evaluated by semi-structured interviews. A semi-structured interview guide will be used to interview the parents and children in the intervention group (aiming 15-30) and healthcare professionals who used ICory-Circumcision. Parents and children will be asked about the contents, activities, and delivery methods, and usefulness of the application. Healthcare professionals will be asked about the strengths and weaknesses of the application and their opinion about the application from their perspective. This is a qualitative data and the data will be analyzed by thematic analysis. Thus, there is no score for this evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Hong-Gu HE, PhD, Principal Investigator — National University of Singapore; Vidyadhar P Mali, PhD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Due to the PDPA in Singapore, PI doesn't plan to share data to public.

REFERENCES:
- [Background] Ahmed MI, Farrell MA, Parrish K, Karla A. Preoperative anxiety in children risk factors and non-pharmacological management. Middle East J Anaesthesiol. 2011 Jun;21(2):153-64. PMID 22435267
- [Background] American Psychiatric Association, & American Psychiatric Association. DSM-5 Task Force. (2013). Diagnostic and statistical manual of mental disorders: DSM-5 (5th ed.). Washington, DC: American Psychiatric Publishing.
- [Background] Arntz A, Dreessen L, De Jong P. The influence of anxiety on pain: attentional and attributional mediators. Pain. 1994 Mar;56(3):307-314. doi: 10.1016/0304-3959(94)90169-4. PMID 8022624
- [Background] Bandura, A. (1997). Self-efficacy: The Exercise of Control. New York: Freeman.
- [Background] Bartik K, Toruner EK. Effectiveness of a Preoperative Preparation Program on Children's Emotional States and Parental Anxiety. J Perianesth Nurs. 2018 Dec;33(6):972-980. doi: 10.1016/j.jopan.2017.09.008. Epub 2017 Nov 20. PMID 30449445
- [Background] Begum, S., Pikkarainen, M., Mali, V.P., Loh, D., Wang, W., & He, H.G.* (2019). Experiences and Needs of Parents following their Child's Paediatric Day Surgery: A Descriptive Qualitative Study. Journal of Pediatric Nursing. (Under preparation)
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Bhansali R, Armstrong J. Smartphone applications for pediatric anesthesia. Paediatr Anaesth. 2012 Apr;22(4):400-4. doi: 10.1111/j.1460-9592.2012.03805.x. Epub 2012 Feb 6. PMID 22309487
- [Background] Björkman, B., Golsäter, M., & Enskär, K. (2014). Children's anxiety, pain, and distress related to the perception of care while undergoing an acute radiographic examination. Journal of Radiology Nursing, 33(2), 69-78. doi:10.1016/j.jradnu.2013.12.003
- [Background] American Academy of Pediatrics Task Force on Circumcision. Circumcision policy statement. Pediatrics. 2012 Sep;130(3):585-6. doi: 10.1542/peds.2012-1989. Epub 2012 Aug 27. PMID 22926180
- [Background] Boker A, Brownell L, Donen N. The Amsterdam preoperative anxiety and information scale provides a simple and reliable measure of preoperative anxiety. Can J Anaesth. 2002 Oct;49(8):792-8. doi: 10.1007/BF03017410. PMID 12374706
- [Background] Bowen, L., & Thomas, M. (2016). Paediatric day case surgery. Anaesthesia and Intensive Care Medicine, 17(6), 274-279. doi:10.1016/j.mpaic.2016.03.008
- [Background] Bradley EH, Curry LA, Devers KJ. Qualitative data analysis for health services research: developing taxonomy, themes, and theory. Health Serv Res. 2007 Aug;42(4):1758-72. doi: 10.1111/j.1475-6773.2006.00684.x. PMID 17286625
- [Background] Braun, V., & Clarke, V. (2006). Using thematic analysis in psychology. Qualitative Research in Psychology, 3(2), 77-101.
- [Background] Tural Buyuk E, Bolisik B. An Analysis of the Anxiety Levels of Mothers Who Participate in Education and Therapeutic Games About Their Children's Surgeries. J Perianesth Nurs. 2018 Jun;33(3):290-295. doi: 10.1016/j.jopan.2016.09.011. Epub 2017 Apr 12. PMID 29784258
- [Background] Capurso M, Ragni B. Psycho-educational preparation of children for anaesthesia: A review of intervention methods. Patient Educ Couns. 2016 Feb;99(2):173-85. doi: 10.1016/j.pec.2015.09.004. Epub 2015 Oct 3. PMID 26603504
- [Background] Chahal N, Manlhiot C, Colapinto K, Van Alphen J, McCrindle BW, Rush J. Association between parental anxiety and compliance with preoperative requirements for pediatric outpatient surgery. J Pediatr Health Care. 2009 Nov-Dec;23(6):372-7. doi: 10.1016/j.pedhc.2008.08.002. Epub 2008 Oct 23. PMID 19875024
- [Background] Chang CM, Li Y, Or LL, Pikkarainen M, Polkki T, Wang W, Lau ST, He HG. A Qualitative Study Exploring Singaporean Parents' Perceptions on PreParing their Child for Surgery. J Pediatr Nurs. 2020 Sep-Oct;54:e69-e77. doi: 10.1016/j.pedn.2020.05.004. Epub 2020 May 27. PMID 32473825
- [Background] Chieng YJ, Chan WC, Klainin-Yobas P, He HG. Perioperative anxiety and postoperative pain in children and adolescents undergoing elective surgical procedures: a quantitative systematic review. J Adv Nurs. 2014 Feb;70(2):243-55. doi: 10.1111/jan.12205. Epub 2013 Jul 19. PMID 23865442
- [Background] Chieng YJ, Chan WC, Liam JL, Klainin-Yobas P, Wang W, He HG. Exploring influencing factors of postoperative pain in school-age children undergoing elective surgery. J Spec Pediatr Nurs. 2013 Jul;18(3):243-52. doi: 10.1111/jspn.12030. Epub 2013 Apr 23. PMID 23822848
- [Background] Chng HY, He HG, Chan SW, Liam JL, Zhu L, Cheng KK. Parents' knowledge, attitudes, use of pain relief methods and satisfaction related to their children's postoperative pain management: a descriptive correlational study. J Clin Nurs. 2015 Jun;24(11-12):1630-42. doi: 10.1111/jocn.12764. Epub 2015 Feb 7. PMID 25661273
- [Background] Chow CH, Van Lieshout RJ, Schmidt LA, Dobson KG, Buckley N. Systematic Review: Audiovisual Interventions for Reducing Preoperative Anxiety in Children Undergoing Elective Surgery. J Pediatr Psychol. 2016 Mar;41(2):182-203. doi: 10.1093/jpepsy/jsv094. Epub 2015 Oct 17. PMID 26476281
- [Background] Cohen LL, Lemanek K, Blount RL, Dahlquist LM, Lim CS, Palermo TM, McKenna KD, Weiss KE. Evidence-based assessment of pediatric pain. J Pediatr Psychol. 2008 Oct;33(9):939-55; discussion 956-7. doi: 10.1093/jpepsy/jsm103. Epub 2007 Nov 17. PMID 18024983
- [Background] Crevatin F, Cozzi G, Braido E, Bertossa G, Rizzitelli P, Lionetti D, Matassi D, Calusa D, Ronfani L, Barbi E. Hand-held computers can help to distract children undergoing painful venipuncture procedures. Acta Paediatr. 2016 Aug;105(8):930-4. doi: 10.1111/apa.13454. Epub 2016 May 23. PMID 27128220
- [Background] Cumino DO, Vieira JE, Lima LC, Stievano LP, Silva RA, Mathias LA. Smartphone-based behavioural intervention alleviates children's anxiety during anaesthesia induction: A randomised controlled trial. Eur J Anaesthesiol. 2017 Mar;34(3):169-175. doi: 10.1097/EJA.0000000000000589. PMID 28146459
- [Background] Cypress BS. Rigor or Reliability and Validity in Qualitative Research: Perspectives, Strategies, Reconceptualization, and Recommendations. Dimens Crit Care Nurs. 2017 Jul/Aug;36(4):253-263. doi: 10.1097/DCC.0000000000000253. PMID 28570380
- [Background] Doig GS, Simpson F. Randomization and allocation concealment: a practical guide for researchers. J Crit Care. 2005 Jun;20(2):187-91; discussion 191-3. doi: 10.1016/j.jcrc.2005.04.005. PMID 16139163
- [Background] Eaton LH, Doorenbos AZ, Schmitz KL, Carpenter KM, McGregor BA. Establishing treatment fidelity in a web-based behavioral intervention study. Nurs Res. 2011 Nov-Dec;60(6):430-5. doi: 10.1097/NNR.0b013e31823386aa. PMID 22048559
- [Background] Fairman, A.D. (2013). Developing self-management skills in persons with spina bifida through mHealth applications: design and clinical efficacy. PhD thesis. University of Pittsburgh.
- [Background] Fortier MA, Del Rosario AM, Martin SR, Kain ZN. Perioperative anxiety in children. Paediatr Anaesth. 2010 Apr;20(4):318-22. doi: 10.1111/j.1460-9592.2010.03263.x. Epub 2010 Feb 23. PMID 20199609
- [Background] Gao, X. L., Liu, Y., Tian, S., Zhang, D. Q., & Wu, Q. P. (2014). Effect of interesting games on relief of preoperative anxiety in preschool children. International Journal of Nursing Sciences, 1(1), 89-92. doi:10.1016/j.ijnss.2014.02.002
- [Background] Goebel S, Mehdorn HM. Assessment of preoperative anxiety in neurosurgical patients: Comparison of widely used measures and recommendations for clinic and research. Clin Neurol Neurosurg. 2018 Sep;172:62-68. doi: 10.1016/j.clineuro.2018.06.036. Epub 2018 Jul 2. PMID 29986197
- [Background] Gubrium, J. F., & Holstein, J. A. (2001). Handbook of interview research. : SAGE Publications, Inc. doi: 10.4135/9781412973588
- [Background] Gilbert, G. E., & Prion, S. (2016). Making sense of methods and measurement: Lawshe's content validity index. Clinical Simulation in Nursing, 12(12), 530-531. doi:10.1016/j.ecns.2016.08.002
- [Background] Hariton E, Locascio JJ. Randomised controlled trials - the gold standard for effectiveness research: Study design: randomised controlled trials. BJOG. 2018 Dec;125(13):1716. doi: 10.1111/1471-0528.15199. Epub 2018 Jun 19. No abstract available. PMID 29916205
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Zhu L, Chan WS, Liam JLW, Xiao C, Lim ECC, Luo N, Cheng KFK, He HG. Effects of postoperative pain management educational interventions on the outcomes of parents and their children who underwent an inpatient elective surgery: A randomized controlled trial. J Adv Nurs. 2018 Jul;74(7):1517-1530. doi: 10.1111/jan.13573. Epub 2018 Apr 23. PMID 29574988
- [Background] He, H. G., Chan, W. C. S., Cheng, K. K. F., Luo, N. Liam, L. W. J., Zhu, L. X., Xiao, C. X., Saw, S. K., & Lim, E. (2013b). Parents' Guide: managing your child's postoperative pain [Video] (English narration, with English, Chinese and Malay subtitles). Singapore: Alice Lee Centre for Nursing Studies, National University of Singapore, and KK Women's and Children's Hospital, Singapore.
- [Background] He, H. G., & Jahja, R. (2008). Postoperative pain management in school-aged children: Emphasis on non-pharmacological methods. Booklet for nurses. Alice Lee Centre for Nursing Studies, National University of Singapore, Singapore.
- [Background] He HG, Jahja R, Lee TL, Ang EN, Sinnappan R, Vehvilainen-Julkunen K, Chan MF. Nurses' use of non-pharmacological methods in children's postoperative pain management: educational intervention study. J Adv Nurs. 2010 Nov;66(11):2398-409. doi: 10.1111/j.1365-2648.2010.05402.x. Epub 2010 Aug 16. PMID 20722797
- [Background] He HG, Jahja R, Sinnappan R, Ang EN, Lee TL, Chan MF, Vehvilainen-Julkunen K. Singaporean nurses' provision of guidance to parents on non-pharmacological postoperative pain-relief methods: An educational intervention study. Nurs Health Sci. 2011 Sep;13(3):344-51. doi: 10.1111/j.1442-2018.2011.00624.x. Epub 2011 Aug 3. PMID 21812878
- [Background] He HG, Klainin-Yobas P, Ang EN, Sinnappan R, Polkki T, Wang W. Nurses' provision of parental guidance regarding school-aged children's postoperative pain management: a descriptive correlational study. Pain Manag Nurs. 2015 Feb;16(1):40-50. doi: 10.1016/j.pmn.2014.03.002. Epub 2014 Jun 21. PMID 24957816
- [Background] He HG, Lee TL, Jahja R, Sinnappan R, Vehvilainen-Julkunen K, Polkki T, Ang EN. The use of nonpharmacological methods for children's postoperative pain relief: Singapore nurses' perspectives. J Spec Pediatr Nurs. 2011 Jan;16(1):27-38. doi: 10.1111/j.1744-6155.2010.00268.x. PMID 21294833
- [Background] He HG, Polkki T, Pietila AM, Vehvilainen-Julkunen K. Chinese parent's use of nonpharmacological methods in children's postoperative pain relief. Scand J Caring Sci. 2006 Mar;20(1):2-9. doi: 10.1111/j.1471-6712.2006.00373.x. PMID 16489954
- [Background] He HG, Polkki T, Vehvilainen-Julkunen K, Pietila AM. Chinese nurses' use of non-pharmacological methods in children's postoperative pain relief. J Adv Nurs. 2005 Aug;51(4):335-42. doi: 10.1111/j.1365-2648.2005.03505.x. PMID 16086802
- [Background] He HG, Polkki T, Pietila AM, Vehvilainen-Julkunen K. A survey of Chinese nurses' guidance to parents in children's postoperative pain relief. J Clin Nurs. 2005 Oct;14(9):1075-82. doi: 10.1111/j.1365-2702.2005.01216.x. PMID 16164525
- [Background] He HG, Vehvilainen-Julkunen K, Pietila AM, Polkki T. Increasing nurses' knowledge and behavior changes in nonpharmacological pain management for children in China. J Nurs Care Qual. 2008 Apr-Jun;23(2):170-6. doi: 10.1097/01.NCQ.0000313767.09891.0a. PMID 18344784
- [Background] He HG, Vehvilainen-Julkunen K, Polkki T, Pietila AM. Children's perceptions on the implementation of methods for their postoperative pain alleviation: an interview study. Int J Nurs Pract. 2007 Apr;13(2):89-99. doi: 10.1111/j.1440-172X.2007.00614.x. PMID 17394516
- [Background] He HG, Vehvilainen-Julkunen K, Polkki T, Pietila AM. Chinese parents' perception of support received and recommendations regarding children's postoperative pain management. Int J Nurs Pract. 2010 Jun;16(3):254-61. doi: 10.1111/j.1440-172X.2010.01838.x. PMID 20618535
- [Background] He HG, Zhu L, Li HC, Wang W, Vehvilainen-Julkunen K, Chan SW. A randomized controlled trial of the effectiveness of a therapeutic play intervention on outcomes of children undergoing inpatient elective surgery: study protocol. J Adv Nurs. 2014 Feb;70(2):431-42. doi: 10.1111/jan.12234. Epub 2013 Aug 29. PMID 23991679
- [Background] He HG, Zhu L, Chan SW, Liam JL, Li HC, Ko SS, Klainin-Yobas P, Wang W. Therapeutic play intervention on children's perioperative anxiety, negative emotional manifestation and postoperative pain: a randomized controlled trial. J Adv Nurs. 2015 May;71(5):1032-43. doi: 10.1111/jan.12608. Epub 2015 Jan 6. PMID 25561079
- [Background] He HG, Zhu LX, Chan WC, Liam JL, Ko SS, Li HC, Wang W, Yobas P. A mixed-method study of effects of a therapeutic play intervention for children on parental anxiety and parents' perceptions of the intervention. J Adv Nurs. 2015 Jul;71(7):1539-51. doi: 10.1111/jan.12623. Epub 2015 Feb 12. PMID 25682703
- [Background] He HG, Zhu L, Chan WC, Xiao C, Klainin-Yobas P, Wang W, Cheng KF, Luo N. A randomized controlled trial of the effectiveness of an educational intervention on outcomes of parents and their children undergoing inpatient elective surgery: study protocol. J Adv Nurs. 2015 Mar;71(3):665-75. doi: 10.1111/jan.12521. Epub 2014 Sep 12. PMID 25212474
- [Background] He HG, Zhu L, Chan SW, Klainin-Yobas P, Wang W. The effectiveness of therapeutic play intervention in reducing perioperative anxiety, negative behaviors, and postoperative pain in children undergoing elective surgery: a systematic review. Pain Manag Nurs. 2015 Jun;16(3):425-39. doi: 10.1016/j.pmn.2014.08.011. PMID 26025800
- [Background] Healy K. A descriptive survey of the information needs of parents of children admitted for same day surgery. J Pediatr Nurs. 2013 Apr;28(2):179-85. doi: 10.1016/j.pedn.2012.07.010. Epub 2012 Aug 11. PMID 22892072
- [Background] Himes MK, Munyer K, Henly SJ. Parental presence during pediatric anesthetic inductions. AANA J. 2003 Aug;71(4):293-8. PMID 13677225
- [Background] Holloway, I., & Wheeler, S. (2002). Qualitative Research in Nursing (2nd edn). Oxford: Blackwell Science Ltd.
- [Background] Hoque R, Sorwar G. Understanding factors influencing the adoption of mHealth by the elderly: An extension of the UTAUT model. Int J Med Inform. 2017 May;101:75-84. doi: 10.1016/j.ijmedinf.2017.02.002. Epub 2017 Feb 10. PMID 28347450
- [Background] Hug M, Tonz M, Kaiser G. Parental stress in paediatric day-case surgery. Pediatr Surg Int. 2005 Feb;21(2):94-9. doi: 10.1007/s00383-004-1333-1. Epub 2005 Jan 5. PMID 15633051
- [Background] Huguet A, Stinson JN, McGrath PJ. Measurement of self-reported pain intensity in children and adolescents. J Psychosom Res. 2010 Apr;68(4):329-36. doi: 10.1016/j.jpsychores.2009.06.003. Epub 2009 Oct 2. PMID 20307699
- [Background] Hui, W. J. (2019). Parental experiences while waiting for children undergoing surgery: A descriptive qualitative study. (Unpublished honours thesis). National University of Singapore, Singapore
- [Background] Hung YC, Chang DC, Westfal ML, Marks IH, Masiakos PT, Kelleher CM. A Longitudinal Population Analysis of Cumulative Risks of Circumcision. J Surg Res. 2019 Jan;233:111-117. doi: 10.1016/j.jss.2018.07.069. Epub 2018 Aug 18. PMID 30502236
- [Background] Jenkins BN, Fortier MA, Kaplan SH, Mayes LC, Kain ZN. Development of a short version of the modified Yale Preoperative Anxiety Scale. Anesth Analg. 2014 Sep;119(3):643-650. doi: 10.1213/ANE.0000000000000350. PMID 25010821
- [Background] Justus R, Wyles D, Wilson J, Rode D, Walther V, Lim-Sulit N. Preparing children and families for surgery: Mount Sinai's multidisciplinary perspective. Pediatr Nurs. 2006 Jan-Feb;32(1):35-43. PMID 16572537
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Karanicolas PJ, Farrokhyar F, Bhandari M. Practical tips for surgical research: blinding: who, what, when, why, how? Can J Surg. 2010 Oct;53(5):345-8. No abstract available. PMID 20858381
- [Background] Kassai B, Rabilloud M, Dantony E, Grousson S, Revol O, Malik S, Ginhoux T, Touil N, Chassard D, Pereira de Souza Neto E. Introduction of a paediatric anaesthesia comic information leaflet reduced preoperative anxiety in children. Br J Anaesth. 2016 Jul;117(1):95-102. doi: 10.1093/bja/aew154. PMID 27317708
- [Background] Kortesluoma RL, Nikkonen M, Serlo W. "You just have to make the pain go away"--children's experiences of pain management. Pain Manag Nurs. 2008 Dec;9(4):143-9, 149.e1-5. doi: 10.1016/j.pmn.2008.07.002. PMID 19041611
- [Background] Kumar A, Das S, Chauhan S, Kiran U, Satapathy S. Perioperative Anxiety and Stress in Children Undergoing Congenital Cardiac Surgery and Their Parents: Effect of Brief Intervention-A Randomized Control Trial. J Cardiothorac Vasc Anesth. 2019 May;33(5):1244-1250. doi: 10.1053/j.jvca.2018.08.187. Epub 2018 Aug 22. PMID 30243867
- [Background] Kushnir J, Djerassi R, Sofer T, Kushnir T. Threat perception, anxiety and noncompliance with preoperative fasting instructions among mothers of children attending elective same day surgery. J Pediatr Surg. 2015 May;50(5):869-74. doi: 10.1016/j.jpedsurg.2014.08.018. Epub 2014 Oct 1. PMID 25783336
- [Background] Lamontagne LL, Hepworth JT, Salisbury MH. Anxiety and postoperative pain in children who undergo major orthopedic surgery. Appl Nurs Res. 2001 Aug;14(3):119-24. doi: 10.1053/apnr.2001.24410. PMID 11481590
- [Background] Lee JH, Jung HK, Lee GG, Kim HY, Park SG, Woo SC. Effect of behavioral intervention using smartphone application for preoperative anxiety in pediatric patients. Korean J Anesthesiol. 2013 Dec;65(6):508-18. doi: 10.4097/kjae.2013.65.6.508. Epub 2013 Dec 26. PMID 24427456
- [Background] Li HC, Lam HY. Paediatric day surgery: impact on Hong Kong Chinese children and their parents. J Clin Nurs. 2003 Nov;12(6):882-7. doi: 10.1046/j.1365-2702.2003.00805.x. PMID 14632981
- [Background] Li HC, Lopez V. The reliability and validity of the Chinese version of the Trait Anxiety Scale for Children. Res Nurs Health. 2004 Dec;27(6):426-34. doi: 10.1002/nur.20045. PMID 15514957
- [Background] Li HC, Lopez V. Children's Emotional Manifestation Scale: development and testing. J Clin Nurs. 2005 Feb;14(2):223-9. doi: 10.1111/j.1365-2702.2004.01031.x. PMID 15669931
- [Background] William Li HC, Lopez V, Lee TL. Effects of preoperative therapeutic play on outcomes of school-age children undergoing day surgery. Res Nurs Health. 2007 Jun;30(3):320-32. doi: 10.1002/nur.20191. PMID 17514706
- [Background] Li HC, Lopez V, Lee TL. Psychoeducational preparation of children for surgery: the importance of parental involvement. Patient Educ Couns. 2007 Jan;65(1):34-41. doi: 10.1016/j.pec.2006.04.009. Epub 2006 Jul 26. PMID 16872785
- [Background] Lim SH, Mackey S, Liam JL, He HG. An exploration of Singaporean parental experiences in managing school-aged children's postoperative pain: a descriptive qualitative approach. J Clin Nurs. 2012 Mar;21(5-6):860-9. doi: 10.1111/j.1365-2702.2011.03911.x. Epub 2011 Nov 15. PMID 22081992
- [Background] Linton, S. J., & Linton, S. (2005). Understanding pain for better clinical practice: A psychological perspective. St. Louis: Elsevier Health Sciences.
- [Background] Longard J, Twycross A, Williams AM, Hong P, Chorney J. Parents' experiences of managing their child's postoperative pain at home: an exploratory qualitative study. J Clin Nurs. 2016 Sep;25(17-18):2619-28. doi: 10.1111/jocn.13307. Epub 2016 Jun 27. PMID 27349504
- [Background] Mali, V. P., Prabhakaran, K., Yee, K. F., Hota, S., Tang, K. P. (2008). Elimination of attendance to children's emergency following circumcision in children. Sustainability award, Clinical Practice Improvement Project. National Healthcare Group, Singapore, 2008.
- [Background] Matthews, J. N. S. (2000). An introduction to randomized controlled clinical trials. London: Arnold; New York: co-published in the U.S. by Oxford University Press.
- [Background] Matthews, J. N. S. (2006). Introduction to randomized controlled clinical trials (2nd ed.). Boca Raton, FL: Chapman & Hall/CRC.
- [Background] Meletti DP, Meletti JFA, Camargo RPS, Silva LM, Modolo NSP. Psychological preparation reduces preoperative anxiety in children. Randomized and double-blind trial. J Pediatr (Rio J). 2019 Sep-Oct;95(5):545-551. doi: 10.1016/j.jped.2018.05.009. Epub 2018 Jun 30. PMID 31340899
- [Background] Mishra P, Foley D, Rutlede E, Allford M. Is day surgery failing our children? J Paediatr Child Health. 2015 Oct;51(10):960-1. doi: 10.1111/jpc.12958. No abstract available. PMID 26428421
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Morris BJ, Wamai RG, Henebeng EB, Tobian AA, Klausner JD, Banerjee J, Hankins CA. Estimation of country-specific and global prevalence of male circumcision. Popul Health Metr. 2016 Mar 1;14:4. doi: 10.1186/s12963-016-0073-5. eCollection 2016. PMID 26933388
- [Background] Munro, B. H. (2005). Statistical Methods for Health Care Research (5th ed.). United States of America: Lippincott Williams & Wilkins.
- [Background] Navaratnarajah, J., & Thomas, M. (2013). Day surgery for children. Anaesthesia and Intensive Care Medicine, 14(6), 232-236. doi:10.1016/j.mpaic.2013.04.015
- [Background] Nilsson S, Enskar K, Hallqvist C, Kokinsky E. Active and passive distraction in children undergoing wound dressings. J Pediatr Nurs. 2013 Apr;28(2):158-66. doi: 10.1016/j.pedn.2012.06.003. Epub 2012 Jul 20. PMID 22819747
- [Background] Patel A, Schieble T, Davidson M, Tran MC, Schoenberg C, Delphin E, Bennett H. Distraction with a hand-held video game reduces pediatric preoperative anxiety. Paediatr Anaesth. 2006 Oct;16(10):1019-27. doi: 10.1111/j.1460-9592.2006.01914.x. PMID 16972829
- [Background] Peterson AM, Harper FW, Albrecht TL, Taub JW, Orom H, Phipps S, Penner LA. Parent caregiver self-efficacy and child reactions to pediatric cancer treatment procedures. J Pediatr Oncol Nurs. 2014 Jan-Feb;31(1):18-27. doi: 10.1177/1043454213514792. Epub 2013 Dec 30. PMID 24378818
- [Background] Pfuntner, A., Wier, L. M., Stocks, C. (2013). Most frequent procedures performed in US hospitals, 2011: Statistical brief# 165. Rockville, MD: Agency for Health Care Policy and Research.
- [Background] Polit, D. F., & Beck, C. T. (2008). Nursing Research: Principles and Methods. (8th ed.). Philadelphia: Lippincott Williams & Wilkins.
- [Background] Power NM, Howard RF, Wade AM, Franck LS. Pain and behaviour changes in children following surgery. Arch Dis Child. 2012 Oct;97(10):879-84. doi: 10.1136/archdischild-2011-301378. Epub 2012 Jul 17. PMID 22806233
- [Background] Pritchard MJ. Identifying and assessing anxiety in pre-operative patients. Nurs Stand. 2009 Aug 26;23(51):35-40. doi: 10.7748/ns.23.51.35.s46. No abstract available. PMID 28075906
- [Background] Rabbitts JA, Groenewald CB, Tai GG, Palermo TM. Presurgical psychosocial predictors of acute postsurgical pain and quality of life in children undergoing major surgery. J Pain. 2015 Mar;16(3):226-34. doi: 10.1016/j.jpain.2014.11.015. Epub 2014 Dec 22. PMID 25540939
- [Background] Radesky JS, Schumacher J, Zuckerman B. Mobile and interactive media use by young children: the good, the bad, and the unknown. Pediatrics. 2015 Jan;135(1):1-3. doi: 10.1542/peds.2014-2251. No abstract available. PMID 25548323
- [Background] Rema, J.P., Cavaleiro, C., Pina, P., Machado, M.S. (2016). Preoperative anxiety in preschool children - observational study. Journal of Anesthesia and Clinical Research. 7(9), 669. doi:10.4172/2155-6148.1000669
- [Background] Robinson EM, Baker R, Hossain MM. Randomized Trial Evaluating the Effectiveness of Coloring on Decreasing Anxiety Among Parents in a Pediatric Surgical Waiting Area. J Pediatr Nurs. 2018 Jul-Aug;41:80-83. doi: 10.1016/j.pedn.2018.02.001. Epub 2018 Feb 10. PMID 29439840
- [Background] Rodriguez S, Caruso T, Tsui B. Bedside Entertainment and Relaxation Theater: size and novelty does matter when using video distraction for perioperative pediatric anxiety. Paediatr Anaesth. 2017 Jun;27(6):668-669. doi: 10.1111/pan.13133. No abstract available. PMID 28474813
- [Background] Rodriguez S, Tsui JH, Jiang SY, Caruso TJ. Interactive video game built for mask induction in pediatric patients. Can J Anaesth. 2017 Oct;64(10):1073-1074. doi: 10.1007/s12630-017-0922-0. Epub 2017 Jun 23. No abstract available. PMID 28646461
- [Background] Sabri, H., Cowan, B., Kapralos, B., Porte, M., Backstein, D., & Dubrowskie, A. (2010). Serious games for knee replacement surgery procedure education and training. Procedia - Social and Behavioral Sciences, 2(2), 3483-3488. doi:10.1016/j.sbspro.2010.03.539
- [Background] Sandelowski M. What's in a name? Qualitative description revisited. Res Nurs Health. 2010 Feb;33(1):77-84. doi: 10.1002/nur.20362. PMID 20014004
- [Background] Schulz KF, Grimes DA. Allocation concealment in randomised trials: defending against deciphering. Lancet. 2002 Feb 16;359(9306):614-8. doi: 10.1016/S0140-6736(02)07750-4. PMID 11867132
- [Background] Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.
- [Background] Seiden SC, McMullan S, Sequera-Ramos L, De Oliveira GS Jr, Roth A, Rosenblatt A, Jesdale BM, Suresh S. Tablet-based Interactive Distraction (TBID) vs oral midazolam to minimize perioperative anxiety in pediatric patients: a noninferiority randomized trial. Paediatr Anaesth. 2014 Dec;24(12):1217-23. doi: 10.1111/pan.12475. Epub 2014 Jul 17. PMID 25040433
- [Background] Sng QW, Taylor B, Liam JL, Klainin-Yobas P, Wang W, He HG. Postoperative pain management experiences among school-aged children: a qualitative study. J Clin Nurs. 2013 Apr;22(7-8):958-68. doi: 10.1111/jocn.12052. Epub 2013 Jan 12. PMID 23311588
- [Background] Sng QW, He HG, Wang W, Taylor B, Chow A, Klainin-Yobas P, Zhu L. A Meta-Synthesis of Children's Experiences of Postoperative Pain Management. Worldviews Evid Based Nurs. 2017 Feb;14(1):46-54. doi: 10.1111/wvn.12185. Epub 2016 Dec 8. PMID 27930859
- [Background] Sobo EJ. Parents' perceptions of pediatric day surgery risks: unforeseeable complications, or avoidable mistakes? Soc Sci Med. 2005 May;60(10):2341-50. doi: 10.1016/j.socscimed.2004.10.006. Epub 2004 Dec 16. PMID 15748681
- [Background] Stanley M, Pollard D. Relationship between knowledge, attitudes, and self-efficacy of nurses in the management of pediatric pain. Pediatr Nurs. 2013 Jul-Aug;39(4):165-71. PMID 24027950
- [Background] Stinson JN, Kavanagh T, Yamada J, Gill N, Stevens B. Systematic review of the psychometric properties, interpretability and feasibility of self-report pain intensity measures for use in clinical trials in children and adolescents. Pain. 2006 Nov;125(1-2):143-57. doi: 10.1016/j.pain.2006.05.006. Epub 2006 Jun 13. PMID 16777328
- [Background] Sun J, Guo Y, Wang X, Zeng Q. mHealth For Aging China: Opportunities and Challenges. Aging Dis. 2016 Jan 2;7(1):53-67. doi: 10.14336/AD.2015.1011. eCollection 2016 Jan. PMID 26816664
- [Background] Sutters KA, Savedra MC, Miaskowski C, Holdridge-Zeuner D, Waite S, Paul SM, Lanier B. Children's expectations of pain, perceptions of analgesic efficacy, and experiences with nonpharmacologic pain management strategies at home following tonsillectomy. J Spec Pediatr Nurs. 2007 Jul;12(3):139-48. doi: 10.1111/j.1744-6155.2007.00107.x. PMID 17594294
- [Background] Taylor, B., Kermode, S., & Roberts, K. (2006). Research in Nursing and Healthcare, 3rd edn. Sydney: Thomson.
- [Background] Upadhyaya, M., & Lander, A. (2013). Day-case surgery in children. Surgery, 31(3), 140-144. doi:10.1016/j.mpsur.2013.01.010
- [Background] Vaughn F, Wichowski H, Bosworth G. Does preoperative anxiety level predict postoperative pain? AORN J. 2007 Mar;85(3):589-604. doi: 10.1016/S0001-2092(07)60130-6. PMID 17352896
- [Background] von Baeyer CL. Children's self-reports of pain intensity: scale selection, limitations and interpretation. Pain Res Manag. 2006 Autumn;11(3):157-62. doi: 10.1155/2006/197616. PMID 16960632
- [Background] Wang W, Zhang H, Lopez V, Wu VX, Poo DC, Kowitlawakul Y. Improving awareness, knowledge and heart-related lifestyle of coronary heart disease among working population through a mHealth programme: study protocol. J Adv Nurs. 2015 Sep;71(9):2200-7. doi: 10.1111/jan.12668. Epub 2015 Apr 16. PMID 25879395
- [Background] Wennstrom B, Tornhage CJ, Hedelin H, Nasic S, Bergh I. Child drawings and salivary cortisol in children undergoing preoperative procedures associated with day surgery. J Perianesth Nurs. 2013 Dec;28(6):361-7. doi: 10.1016/j.jopan.2013.05.009. PMID 24267624
- [Background] Wong, G. G. (2018). Preliminary effects of using mobile games to reduce perioperative anxiety and postoperative pain in children undergoing elective surgery: A mixed methods study. (Unpublished honours thesis). National University of Singapore, Singapore.
- [Background] Wright KD, Raazi M, Walker KL. Internet-delivered, preoperative, preparation program (I-PPP): Development and examination of effectiveness. J Clin Anesth. 2017 Jun;39:45-52. doi: 10.1016/j.jclinane.2017.03.007. Epub 2017 Mar 27. PMID 28494907
- [Background] Yun OB, Kim SJ, Jung D. Effects of a Clown-Nurse Educational Intervention on the Reduction of Postoperative Anxiety and Pain Among Preschool Children and Their Accompanying Parents in South Korea. J Pediatr Nurs. 2015 Nov-Dec;30(6):e89-99. doi: 10.1016/j.pedn.2015.03.003. Epub 2015 Apr 13. PMID 25882469
- [Background] Ziegler DB, Prior MM. Preparation for surgery and adjustment to hospitalization. Nurs Clin North Am. 1994 Dec;29(4):655-69. PMID 7527524
- [Derived] Kwa ZY, Li J, Loh DL, Lee YY, Liu G, Zhu L, Pikkarainen M, He H, Mali VP. An Intelligent Customer-Driven Digital Solution to Improve Perioperative Health Outcomes Among Children Undergoing Circumcision and Their Parents: Development and Evaluation. JMIR Form Res. 2024 Feb 16;8:e52337. doi: 10.2196/52337. PMID 38363589
- See also: Singapore census of population 2010, statistical release 1: Demographic characteristics, education, language and religion. — https://www.singstat.gov.sg/publications/cop2010/census10_stat_release1
- See also: Statistics on telecom services for 2017 (Jan-Jun) — https://www.imda.gov.sg/industry-development/facts-and-figures/telecommunications/statistics-on-telecom-services/statistic-on-telecom-service-for-2017-jan
- See also: Faces pain scale - revised home — https://www.iasp-pain.org/Education/Content.aspx?ItemNumber=1519&navItemNumber=577
- See also: Buddy Healthcare joining the ICory project. Buddy Healthcare — https://www.buddyhealthcare.com/news/buddy-healthcare-icory-project
- See also: Research Electronic Data Capture — https://projectredcap.org/
- See also: Research Randomizer — https://www.randomizer.org/
- See also: State-Trait Anxiety Inventory (STAI): Mind Garden — https://www.mindgarden.com/146-state-trait-anxiety-inventory-for-children
- See also: Play is the way to healthier life. — https://triumf.health/news/2018-12-triumf-research